CLINICAL TRIAL: NCT06279052
Title: What Projections Towards the Future During a Period of Transition? A Qualitative Study of Adolescents With Prader-Willi Syndrome
Brief Title: Adolescent Projections During Transition in Prader-Willi Syndrome
Acronym: APT-WILL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/23/0535
Record Dates: First submitted 2024-02-14; First posted 2024-02-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phone interview (Experimental): Patients will then be contacted by the investigator to arrange a telephone appointment date.
  On the day of the telephone appointment, the psychiatry intern will call the patient to conduct the interview which will last between 30 and 60 minutes.
  At the end of the telephone interview, the patient's participation in the research will end.
  Interventions: Behavioral: Phone interview

INTERVENTIONS:
Behavioral: Phone interview — Phone interview during which the experience of the transition to adulthood among adolescents and young adults with Prader Willi Syndrome will be retrieved

SUMMARY:
Single-center, cross-sectional qualitative study seeking to collect the experience of adolescence and the transition to adulthood of people affected by Prader-Willi syndrome in a population. To do this, the present will carry out a qualitative study with a reflexive thematic analysis of the data collected through semi-structured interviews using an interview guide.

ELIGIBILITY:
Inclusion Criteria:

* Patients with genetically confirmed Prader-Willi syndrome
* Patients affiliated or beneficiaries of a social security system
* Patients known and followed by the reference center, presenting sufficient intellectual skills to answer the interview questions

Exclusion Criteria:

* Refusal of family participation (if minor)
* Refusal of participation by the patient or his guardian (if of legal age)

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Experience of the disease and aspirations regarding the future | 1 hour
  The main objective of this study is to explore their experience of the disease and their aspirations regarding their future in a population of older adolescents and young adults with Prader-Willi syndrome. A questionnaire created by the clinical investigator containing personal questions will be applied to all patients. There is no scale.

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire BENVEGNU, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No